CLINICAL TRIAL: NCT03357146
Title: Optical Coherence Tomography Angiography Examinations in Chronic Retinal Artery Occlusion
Acronym: RAO-OCTA
Status: Completed | Type: Observational
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Miklos Schneider MD, PhD, Assistant Professor, Semmelweis University
Other Study IDs: RAO-OCTA-1253
Record Dates: First submitted 2017-11-23; First posted 2017-11-29 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Retinal Artery Occlusion
MeSH Terms: conditions — Retinal Artery Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- CRA: Patients with chronic retinal artery occlusion
  Interventions: Device: Optical coherence tomography angiography
- Control: Healthy
  Interventions: Device: Optical coherence tomography angiography

INTERVENTIONS:
Device: Optical coherence tomography angiography — OCTA scans per built-in device protocol

SUMMARY:
Purpose of the study is to examine the retinal blood flow in chronic cases of retinal artery occlusion with non-invasive, non-contact optical coherence tomography angiography.

DETAILED DESCRIPTION:
Occlusion of the retinal arteries is an emergency which causes sudden, painless unilateral vision loss. Loss of blood flow causes ischemic damage to the retina. The extent of damage depends on the area affected.

Following the acute phase of the disease re-canalization occurs and lesser blood flow can be detected usually without functional recovery.

Purpose of the study is to examine the retinal blood flow in chronic cases of retinal artery occlusion.

Standard procedures to examine this disease include retinoscopy following pupil dilation, fluorescein angiography and more recently, optical coherence tomography (OCT).

The latest direction in OCT development was OCT angiography (OCTA) which is a software upgrade that allows detection of blood flow based on motion contrast. Similar to previous OCT machines OCTA is also non-invasive and non-contact and does not require any intravenous agents.

OCT machines are approved in the EU and the US and are not experimental devices.

The device used in this study is the commercially available Zeiss Cirrus HD OCT Angioplex 5000 that operates with spectral-domain technology.

ELIGIBILITY:
Inclusion Criteria:

* central or branch retinal artery occlusion
* at least 6 months of onset
* signed informed consent

Exclusion Criteria:

* known epilepsy
* incapacity
* presence of optical media opacities that would disturb the imaging
* presence of other retinal diseases that would disturb the evaluation of images

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: White caucasias
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Capillary density in relation to healthy subjects | Through study completion, 1 year

SECONDARY OUTCOMES:
Correlation of capillary density and retinal thickness | Through study completion, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Miklos Schneider, Principal Investigator — Semmelweis University, Department of Ophthalmology
Locations (1):
- Semmelweis University, Department of Ophthalmology, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bonini Filho MA, Adhi M, de Carlo TE, Ferrara D, Baumal CR, Witkin AJ, Reichel E, Kuehlewein L, Sadda SR, Sarraf D, Duker JS, Waheed NK. OPTICAL COHERENCE TOMOGRAPHY ANGIOGRAPHY IN RETINAL ARTERY OCCLUSION. Retina. 2015 Nov;35(11):2339-46. doi: 10.1097/IAE.0000000000000850. PMID 26457398
- [Background] Chalam KV, Sambhav K. Optical Coherence Tomography Angiography in Retinal Diseases. J Ophthalmic Vis Res. 2016 Jan-Mar;11(1):84-92. doi: 10.4103/2008-322X.180709. PMID 27195091
- [Background] Jia Y, Bailey ST, Hwang TS, McClintic SM, Gao SS, Pennesi ME, Flaxel CJ, Lauer AK, Wilson DJ, Hornegger J, Fujimoto JG, Huang D. Quantitative optical coherence tomography angiography of vascular abnormalities in the living human eye. Proc Natl Acad Sci U S A. 2015 May 5;112(18):E2395-402. doi: 10.1073/pnas.1500185112. Epub 2015 Apr 20. PMID 25897021
- [Background] Samara WA, Say EA, Khoo CT, Higgins TP, Magrath G, Ferenczy S, Shields CL. CORRELATION OF FOVEAL AVASCULAR ZONE SIZE WITH FOVEAL MORPHOLOGY IN NORMAL EYES USING OPTICAL COHERENCE TOMOGRAPHY ANGIOGRAPHY. Retina. 2015 Nov;35(11):2188-95. doi: 10.1097/IAE.0000000000000847. PMID 26469536
- [Background] Savastano MC, Lumbroso B, Rispoli M. IN VIVO CHARACTERIZATION OF RETINAL VASCULARIZATION MORPHOLOGY USING OPTICAL COHERENCE TOMOGRAPHY ANGIOGRAPHY. Retina. 2015 Nov;35(11):2196-203. doi: 10.1097/IAE.0000000000000635. PMID 25932558
- [Background] Spaide RF. VOLUME-RENDERED ANGIOGRAPHIC AND STRUCTURAL OPTICAL COHERENCE TOMOGRAPHY. Retina. 2015 Nov;35(11):2181-7. doi: 10.1097/IAE.0000000000000764. PMID 26428608
- [Background] Yu S, Lu J, Cao D, Liu R, Liu B, Li T, Luo Y, Lu L. The role of optical coherence tomography angiography in fundus vascular abnormalities. BMC Ophthalmol. 2016 Jul 13;16:107. doi: 10.1186/s12886-016-0277-2. PMID 27412442